CLINICAL TRIAL: NCT01326858
Title: A Randomized, Double-Masked, Crossover Study to Evaluate the Safety and Comfort of AL-4943A Ophthalmic Solution, 0.7%
Brief Title: Safety and Comfort of AL-4943A Ophthalmic Solution
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: C-10-127
Record Dates: First submitted 2011-03-30; First posted 2011-03-31 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-02

CONDITIONS: Allergic Conjunctivitis
Keywords: Ocular discomfort; AL-4943A Ophthalmic Solution
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Olopatadine Hydrochloride; ketotifen fumarate ophthalmic solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Olopatadine, 0.7% (Experimental): Olopatadine hydrochloride ophthalmic solution, 0.7%, 1 drop instilled in each eye, 1 dose, in Period 1, followed by olopatadine hydrochloride ophthalmic vehicle and ketotifen fumarate ophthalmic solution, 0.025%, Periods 2 and 3, as randomized
  Interventions: Drug: Olopatadine hydrochloride ophthalmic solution, 0.7%; Drug: Olopatadine hydrochloride ophthalmic solution vehicle; Drug: Ketotifen fumarate ophthalmic solution, 0.025%
- Vehicle (Placebo Comparator): Olopatadine hydrochloride ophthalmic solution vehicle, 1 drop instilled in each eye, 1 dose, in Period 1, followed by olopatadine hydrochloride ophthalmic solution, 0.7% and ketotifen fumarate ophthalmic solution, 0.025%, Periods 2 and 3, as randomized
  Interventions: Drug: Olopatadine hydrochloride ophthalmic solution, 0.7%; Drug: Olopatadine hydrochloride ophthalmic solution vehicle; Drug: Ketotifen fumarate ophthalmic solution, 0.025%
- Zaditor (Active Comparator): Ketotifen fumarate ophthalmic solution, 0.025%, 1 drop instilled in each eye, 1 dose, in Period 1, followed by olopatadine hydrochloride ophthalmic solution, 0.7% and olopatadine hydrochloride ophthalmic solution vehicle, Periods 2 and 3, as randomized
  Interventions: Drug: Olopatadine hydrochloride ophthalmic solution, 0.7%; Drug: Olopatadine hydrochloride ophthalmic solution vehicle; Drug: Ketotifen fumarate ophthalmic solution, 0.025%

INTERVENTIONS:
Drug: Olopatadine hydrochloride ophthalmic solution, 0.7% — Treatment A
  Other Names: AL-4943A
Drug: Olopatadine hydrochloride ophthalmic solution vehicle — Treatment B, inactive ingredients used as placebo
Drug: Ketotifen fumarate ophthalmic solution, 0.025% — Treatment C
  Other Names: Zaditor®

SUMMARY:
The purpose of this study is to assess the ocular comfort and safety of olopatadine hydrochloride opthalmic solution. 0.7%.

DETAILED DESCRIPTION:
In this 3-treatment, 3-period, 6-sequence crossover study, each subject will receive all 3 products in randomized order, 1 product at a time, with a washout period of 24 hours between treatment periods. Following instillation of study medication, subjects will complete a 3-minute discomfort profile.

ELIGIBILITY:
Inclusion Criteria:

* Able to be dosed in both eyes, to follow instructions, and willing and able to attend required study visits.
* Negative urine pregnancy test if female of childbearing potential and use adequate birth control throughout the study period.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* History or clinical evidence of ocular herpes simplex or ocular herpes zoster infectious disease.
* History of any clinically significant external ocular disease within 30 days of the start of the study.
* Presence of active blepharitis, active meibomian gland dysfunction, active rosacea affecting the ocular surface/lid margin, active or chronic follicular conjunctivitis, preauricular adenopathy, or any other ocular or periocular abnormality that may affect the study outcomes.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Peak discomfort score over a 3-minute period after drop instillation | Up to Day 3
  Ocular discomfort as measured by Visual Analog Scale (VAS) with 0=none to 50=severe, was assessed by subjects every 30 seconds between 0 to 180 seconds after drop instillation (at 0, 30, 60, 90, 120, 150, and 180 seconds). Peak discomfort (maximum observed VAS discomfort score over the 3-minute period) for each subject in each period was analyzed.

SECONDARY OUTCOMES:
Ocular Symptoms | Up to Day 3
  Ocular symptoms (burning, stinging, tearing, blurring, and stickiness) assessed by the subject after instillation of drop as a single score where 0=none to 9=severe.
Product Acceptability | Up to Day 3
  Product Acceptability assessed by the subject after instillation of drop as a single score where 0=very acceptable and 100=not acceptable.

CONTACTS AND LOCATIONS:
Overall Officials: Abhijit Narvekar, MS, MBBS, Study Director — Alcon Research